CLINICAL TRIAL: NCT00858715
Title: Resistance to Antithrombotic Therapy in Patients Undergoing Angioplasty and Stenting for Cardiovascular Disease - Vienna REACT
Brief Title: Resistance to Antithrombotic Therapy
Acronym: Vienna REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christoph W. Kopp, Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vienna REACT
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Atherosclerosis; Angioplasty
Keywords: Clopidogrel; Aspirin; Antithrombotic therapy; Platelet function testing
MeSH Terms: conditions — Atherosclerosis | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 75 mg clopidogrel + 100 mg aspirin
  Interventions: Drug: aspirin; Drug: clopidogrel
- 2 (Active Comparator): 150 mg clopidogrel + 100 mg aspirin
  Interventions: Drug: aspirin; Drug: clopidogrel

INTERVENTIONS:
Drug: aspirin — 100 mg aspirin
Drug: clopidogrel — 75 mg (Arm 1) and 150 mg (Arm 2)

SUMMARY:
Clopidogrel plays a pivotal role in the antithrombotic regimen after percutaneous intervention with stent implantation. However, response to clopidogrel shows a wide interindividual variability and a high on-treatment residual ADP-inducible platelet reactivity has already been associated with an increased risk for adverse events after coronary stenting. In the present study, platelet reactivity will be determined by 6 different platelet function tests in patients on dual antiplatelet therapy after angioplasty and stenting for peripheral, coronary and carotid artery disease. One hundred patients showing high on-treatment residual ADP-inducible platelet reactivity in 2 or more tests will be randomized to receive either 75mg or 150mg of daily clopidogrel in addition to aspirin for 3 months. The aim of the present study is to investigate the effects of intensified antithrombotic therapy (150mg clopidogrel + 100mg aspirin daily) versus standard antithrombotic therapy (75mg clopidogrel + 100mg aspirin daily) in patients with decreased clopidogrel-mediated platelet inhibition after percutaneous intervention with stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* angioplasty and stenting for peripheral, coronary or carotid artery disease

Exclusion Criteria:

* known aspirin or clopidogrel intolerance
* therapy with vitamin K antagonists (warfarin, phenprocoumon, acenocoumarol)
* treatment with ticlopidine, dipyridamol or nonsteroidal antiinflammatory drugs
* family or personal history of bleeding disorders
* malignant paraproteinemias
* myeloproliferative disorders
* heparin-induced thrombocytopenia
* severe hepatic failure
* known qualitative defects in thrombocyte function
* major surgical procedure within one week before enrollment
* platelet count < 100.000 or > 450.000/µl
* hemoglobin < 8 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Occurence of major adverse cardiovascular events (MACE) | 3 months
Occurence of major adverse cardiovascular events (MACE) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph W. Kopp, M.D., Principal Investigator — Division of Angiology/ Department of Internal Medicine II/ Medical University of Vienna
Locations (1):
- Division of Angiology, Department of Internal Medicine II, Medical University of Vienna, Vienna, Austria